CLINICAL TRIAL: NCT03944551
Title: Use of Bubble Continuous Positive Airway Pressure (bCPAP) With High Flow Settings in Treatment of Respiratory Distress Secondary to Signs of Severe Pneumonia in Pediatric Patients in Mali
Brief Title: Bubble Continuous Positive Airway Pressure for Children With Severe Pneumonia in Mali, Africa
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participant mortality rates were higher than expected.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Center for Vaccine Development - Mali (Other)
Responsible Party: Principal Investigator, Adnan Bhutta, Division Head, Department of Pediatrics, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-82800
Record Dates: First submitted 2019-04-22; First posted 2019-05-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is an unblinded, age-stratified, randomized trial with a 2:1 allocation ratio.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bubble CPAP (Experimental)
  Interventions: Device: Bubble CPAP
- Standard Therapy (Other)
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Device: Bubble CPAP — Those assigned to the bCPAP group will receive a Total flow oxygen at a rate of 2 liters per kilogram to a maximum of 10 liters per minute using the appropriate nasal prongs for the age and size of the patient. The positive end-expiratory pressure (PEEP) provide by bCPAP will start at 8cm HO2. The FIO2 will be adjusted to obtain a saturation of oxygen of 90% or greater.
  Arms: Bubble CPAP
Other: Standard Therapy — For patients in the standard therapy group, oxygen will be delivery by nasal cannula at a flow rate of 4 Liters per minute. If a patient in the standard group after 1 hour of treatment still has a SpO2 < 90% or meeting criteria of treatment failure the patient will be move from the standard therapy group to the bCPAP group.
  Arms: Standard Therapy

SUMMARY:
This study is being conducted in Mali, Africa.

Pneumonia is a respiratory infection of the lungs caused by bacteria or virus. Some children can develop signs of severe pneumonia and as a result, have difficulty breathing and low levels of oxygen in the blood. In some cases this can progress to death. Patients with signs of severe pneumonia require admission to the hospital for treatment and the treatment includes delivery of oxygen. Currently, in the hospital, oxygen is available for delivery by nasal cannula to children. In this case, oxygen is given through a small plastic tube which delivers oxygen through the nose. However, the amount of oxygen that can be given is limited because of the size of the tube and the amount of oxygen that can go through. However, a new device known as the bubble CPAP machine delivers oxygen through the nose in a way that helps the airways to stay open. This is known to provide better support to children less than 1 year of age who have difficulty breathing with signs of severe pneumonia. The purpose of this study is to evaluate the effectiveness of bubble CPAP in Children up to 5 years of age with with signs of severe pneumonia.

DETAILED DESCRIPTION:
This study includes two cohorts. One cohort will participate in an interventional clinical trial and the other cohort will participate in an observational study.

Interventional Cohort:

The first cohort will include 600 children with signs of severe pneumonia, 1 year up to 5 years of age. Signs of severe pneumonia include fast breathing, difficulty breathing and who are very sick (not able to drink, vomiting, having seizures, are very sleepy or with severe malnutrition). Two out of every three children will receive oxygen with the bubble CPAP and one out of every three children will receive treatment with oxygen with regular nasal cannula. The treatment assignment will be determined randomly. We will follow up participants during their entire hospitalization. During this time we will collect information on the child's illness, test results and treatment.

Observational Cohort:

The second cohort will include 450 children with signs of severe pneumonia, under 1 year of age. In Mali, bubble CPAP is currently given as standard of care (when possible) for children with signs of severe pneumonia, under 1 year of age; therefore, children in this cohort will already be receiving bubble CPAP as standard of care prior to enrollment. The only research activities will be to follow the children during their hospitalization and collect information about their clinical condition, test results, treatment and the amount of oxygen required during the hospital admission.

The remainder of the information in this ClinicalTrials.gov registration will refer only to the Intervention Cohort.

ELIGIBILITY:
Inclusion criteria:

Cases must meet the all following inclusion criteria for eligibility to be placed on bCPAP

* Hospitalization
* Age 12 months up to 5 years
* Fast breathing defined as: (Using a timing device to count rate for one full minute)

  * ≥ 40 breath/min in a child aged 12-23 months
  * ≥ 30 breaths/min in a child aged 2-5 years
* Any of the following respiratory signs: wheezing, nasal flaring, chest indrawing, cyanosis, grunting, head nodding, stridor and/or oxygen saturation <90%.
* Informed written consent obtained Or
* Age 12 months up to 5 years
* Weight up to 20Kg
* With cough AND/OR any sign of difficult breathing Plus ONE general danger sign as follow:

  * Not able to drink
  * Persistent vomiting
  * Convulsions
  * Lethargy or unconscious
  * Stridor in a calm child or
  * Severe malnutrition
* Informed written consent obtained

Patients with the following conditions who meet eligible criteria can benefit from bCPAP:

* Bronchiolitis
* Respiratory viral infection
* Lung collapse / atelectasis
* Asthma exacerbation
* Patients with congenital heart disease with heart failure
* Malaria
* Severe Anemia
* Sepsis
* Meningitis
* Any patient with increased respiratory effort who meet the eligible criteria

We will include patients with progression to severe pneumonia during the hospitalization and those ones with chronic diseases too.

Definitions:

* Head nodding: a movement of the head synchronous with inspiration indicating severe respiratory distress
* Chest indrawing: lower chest wall goes in when the child breathes in
* Lethargy: is defined as "an infant who does not wake up on stimulation or, on waking, subsequently moves only on stimulation or does not move at all"
* Not able to drink: refers to "difficulty feeding or not feeding well (in an infant who was previously feeding well)"
* Convulsions: During the enrollment process, the danger sign for 'convulsions' will be collected by asking about the number and duration of seizures.
* Severe malnutrition Severe acute malnutrition is defined as per WHO as the presence of edema of both feet or severe wasting (weight-for-height/length <-3SD) or mid upper arm circumference < 115 mm [19]
* Progression to case definition during hospitalization: Cases that progress to severe pneumonia or meet the inclusion criteria previously mentioned during hospitalization but do not meet the definition during the time of admission because the disease is in the early stages of illness will be included.
* Chronic disease: Children with chronic lung or respiratory disease may be admitted to the study. We will not exclude patients from the study on the basis of a long history of symptoms.

Exclusion criteria:

Cases that meet any of the following exclusion criteria will be ineligible to enroll:

* Skin breakdown around the nose and mouth
* Facial trauma
* Persistent episodes of vomiting: more than 3 episodes in 1 hour.

Ages: 12 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Treatment failure rate | 2 hours
  We define treatment failure as the occurrence of any two or more of the following clinical criteria 2 hour after initiation of an intervention:
  * Severe hypoxemia (Saturation of oxygen SpO2 <85%) after being on one of the study groups treatments for 2 hours
  * Increased in respiratory rate by any amount or if respiratory rate remains unchanged after initiation of treatment as follow:
    * ≥ 40 breath/min in a child aged 12-23 months
    * ≥ 30 breaths/min in a child aged 2-5 years
  * Signs of persistent severe respiratory distress defined as head nodding, severe chest indrawing, stridor, apnea, nasal flaring and or grunting.
  * Dies while in the hospital.

SECONDARY OUTCOMES:
Mortality rate | Through hospital discharge, an average of 1 week
  The difference in mortality between the standard therapy group vs bCPAP group at the time of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan T Bhutta, MBBS, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Center for Vaccine Development - Mali, Bamako, Mali